CLINICAL TRIAL: NCT04666844
Title: Predicting Transfers to Hemodialysis in Peritoneal Dialysis Patients Using the Surprise Question
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Principal Investigator, Wael Hussein, MBBS, Senior Director of Clinical Research, Satellite Healthcare
Other Study IDs: SIH126_PD Suprise Question
Record Dates: First submitted 2020-11-16; First posted 2020-12-14 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Peritoneal Dialysis
Keywords: Surprise Question

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey: Clinicians will be asked to provide responses to the two surprise questions for each of their PD patients.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Observational Study

SUMMARY:
The investigators will assess the prediction performance of the modified Surprise Question (Will the participant be surprised if this patient transfers to hemodialysis in the next 6 months?) for identification of peritoneal dialysis at high risk of transfer to hemodialysis. The investigators will also assess the prediction performance of a modified mortality surprise question (Will the participant be surprised if this patient dies in the next 6 months?).

DETAILED DESCRIPTION:
Physicians and nurses will be asked two questions regarding each of their peritoneal dialysis patients:

1. Will the participant be surprised if this patient transfers to hemodialysis in the next 6 months?
2. Will the participant be surprised if this patient dies in the next 6 months?

Patients will be followed for 6 months for outcomes (with two extra months for ascertainment of outcomes).

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Incident and prevalent PD population at Satellite Healthcare

Exclusion Criteria:

* Age < 18 years
* Patients already enrolled in hospice
* Patients on PD training
* Patients on backup hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients on peritoneal dialysis receiving care at Satellite Healthcare facilities.
Sampling Method: Non-Probability Sample
Enrollment: 2019 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Performance measures of the modified surprise question answered by the physicians as a prediction instrument for transfer to hemodialysis of peritoneal dialysis patients in 6 months. | at 6 months

SECONDARY OUTCOMES:
Performance measures of the modified SQ Responses of the nurses to predict Transfers to hemodialysis | at 6 months
Performance measures of the mortality SQ Responses of the physician and nurses to predict death | at 6 months
Performance of prediction model for transfer to HD developed from variables obtained at baseline. | at 0 months
Comparison of performance of baseline variables model to performance of the SQ model, and to a model that combines baseline variables and the SQ. | at 6 month
Rate of hospitalizations in patients identified as high risk by the surprise question. | at 6 months
Rate of peritonitis in patients identified as high risk by the surprise question. | at 6 months
Proportion of patients identified as high risk who transition to HD. | At time of transfer to hemodialysis, for those who transfer to hemodialysis within the observation period, which is 6 months from response to the surprise question
Proportion of patients who transition to HD who (i) start Home HD and those who (ii) start HD with AVF/AVG - in the whole group and among those identified high or low risk by the surprise question. | At time of transfer to hemodialysis, for those who transfer to hemodialysis within the observation period, which is 6 months from response to the surprise question
Evaluating the agreement of assessments made by the primary nephrologist and the primary nurse of the patient | at baseline
Factors associated with predictions made by the MD and nurse. | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wael Hussein, Principal Investigator — Satellite Healthcare
Locations (1):
- Satellite Healthcare Inc, San Jose, California, United States